CLINICAL TRIAL: NCT03894917
Title: Characterizing Disease Biology, Treatment Patterns and Toxicity in Older Adults With Advanced Hepatocellular Carcinoma
Brief Title: Characterizing Disease Biology, Treatment and Toxicity in Older Adults With Hepatocellular Carcinoma
Status: Recruiting | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Other Study IDs: CTMS 19-0010; HSC20190202H (Other: University of Texas Health Science Center- San Antonio)
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Geriatric Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Participants 65 years or older
  Interventions: Other: Comprehensive Geriatric Assessment (CGA)
- Group 2: Participants less than 65 years

INTERVENTIONS:
Other: Comprehensive Geriatric Assessment (CGA) — Assessments will be done for participants that are 65 years or older.
  Groups: Group 1

SUMMARY:
This is an observational, prospective cohort study that will recruit a diverse sample of 84 participants with newly diagnosed with unresectable, advanced hepatocellular carcinoma (HCC) at the UT Health Cancer Center in San Antonio. This study uses geriatric assessment tools with participants 65 years and older and collects adverse events and exploratory markers of aging for all participants.

DETAILED DESCRIPTION:
The results from this study will allow us to identify unique disease characteristics of older participants and to study treatment patterns that may be barriers to treatment and risk factors for increased morbidity. Characteristics of Comprehensive Geriatric Assessment will be obtained prior to standard interventional treatment for participants that are 65 years or older. Observations will be made of treatment toxicities and cellular senescence with treatment outcomes. Findings from this study will result in the development of R01 intervention studies that develop and validate a treatment algorithm based on these associations to provide older adults with a personalized treatment plan.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or radiographically (CT or MRI) confirmed newly diagnosed hepatocellular carcinoma.
* Age 18 years and older.
* Patients with advanced, unresectable HCC as determined by the treating physician.

Exclusion Criteria:

* Patients with resectable HCC who are still candidates for locoregional therapy
* Patients receiving prior systemic or locoregional therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed with advanced hepatocellular carcinoma (HCC) that cannot be removed with surgery.
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2019-09-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Characterize the Change in disease and treatment patterns of advanced hepatocellular carcinoma (HCC) in older patients in the US. | will be collected at time points: at screening, Month 1, Month 2, Month 4, Month 6, Month 8, Month 10 and Month 12.
  Collection of the participants disease characteristics, clinical and treatment data. Comprehensive geriatrics assessments will be done using bilingual assessments in English and Spanish.

CONTACTS AND LOCATIONS:
Overall Officials: Sukeshi Patel Arora, MD, Principal Investigator — Mays Cancer Center
Locations (1):
- Mays Cancer Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No